CLINICAL TRIAL: NCT06828523
Title: Assessing Perceptual Effects of Interactive Tasks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ji Min Lee, Ph.D., Associate Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00024154-2; R01DC021714 (NIH)
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Listeners will hear recorded speech of PALS and age-matched speakers and indicate what they heard. Recorded speech consists of vowels and consonants produced in non-interactive and interactive tasks. The perceptual judgements will be compared to see whether interactive contexts have similar perceptual effects across the two groups.
  Plans for Assignment - This is a single group study in which all participants will engage in the same tasks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Listener Perception of Speech Produced in Different Task Settings (Experimental): Listeners will hear recorded speech of PALS and age-matched speakers produced within interactive and non-interactive contexts and indicate what they heard.
  Interventions: Behavioral: Listener judgements of speech produced in different tasks

INTERVENTIONS:
Behavioral: Listener judgements of speech produced in different tasks — Listeners will hear recorded speech of PALS and age-matched speakers across interactive and non-interactive tasks and indicate what they heard by clicking one of four words displayed on the screen. Standard attention checks and minimum performance thresholds (Theodore, 2021) will be used to ensure that listeners are engaged and are able to provide meaningful perceptual judgments.

SUMMARY:
In this study, we will evaluate how solo, naive listeners perceive the speech of people with amyotrophic lateral sclerosis (ALS) and age-matched speakers produced across interactive and non-interactive contexts with an unfamiliar, naive interlocutor.

DETAILED DESCRIPTION:
Listeners will hear recorded speech of PALS and age-matched speakers and indicate what they heard. Recorded speech consists of vowels and consonants produced in non-interactive and interactive tasks. The perceptual judgements will be compared to see whether interactive contexts have similar perceptual effects across the two groups.

Plans for Assignment - This is a single group study in which all participants will engage in the same tasks.

Delivery of Intervention: Solo listeners will participate in this study in a remote, asynchronous format. They will be recruited using the online participant recruitment platform Prolific © and will use their own laptop/computer and headphones.

Adequacy of Sample size: We will use n = 1300 listeners to achieve 80% power at alpha of .05 to detect between group differences with the assumption of medium effect sizes (Cohen's f = 0.3).

Adequacy of Analyses: The proposed statistical analyses (Generalized mixed effects regressions) are standard and will be used to analyze the effect of the intervention on the outcome measures described below.

ELIGIBILITY:
Inclusion Criteria:

* passing the remote hearing screening
* having no known speech, language or neurological disorders per self-report
* being a native monolingual speaker of American English
* having no experience communicating with people with dysarthria
* being between the ages of 18 and 65.

Exclusion Criteria:

* None - if volunteer meets the inclusion criteria, then they will be enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Intelligibility of recorded speech | one 20 minute session
  Perceptual judgments will be provided by solo, naïve listeners who did not participate in the interactions. Listeners will hear recorded speech of PALS and age-matched speakers recorded across the different tasks and indicate what they heard. The score will be expressed in percent. The possible range is between 0-100%. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jimin Lee, Ph.D., Principal Investigator — The Pennsylvania State University; Navin Viswanathan, Ph.D., Principal Investigator — The Pennsylvania State University; Anne Olmstead, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Speech Core, Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The project will involve the collection of perceptual judgments and questionnaire data. All deidentified data will be shared through the Open Science Framework (osf.io). All scripts, protocols, procedures, and analyses will be shared along with the deidentified data to ensure that other researchers can verify and build on the presented results. All shared data will be made available in a format that is accessible by open-access software (e.g., R, Open Office, pdf reader). In addition, platform-specific scripts (e.g., experimental software LabVanced) will be shared with explanations so that they may be implemented across different software environments.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after publication of the study.
Access Criteria: All deidentified data, metadata, and related tools will be freely available via Open Science Framework (OSF). The original audio files will be made available (for participants who consent) by request from researchers in the field to ensure responsible use.

REFERENCES:
- [Background] Olmstead, A. J., Viswanathan, N., Cowan, T., & Yang, K. (2021). Phonetic adaptation in interlocutors with mismatched language backgrounds: A case for a phonetic synergy account. Journal of Phonetics, 87, 101054. . : . .
- [Background] Olmstead AJ, Lee J, Viswanathan N. The Role of the Speaker, the Listener, and Their Joint Contributions During Communicative Interactions: A Tripartite View of Intelligibility in Individuals With Dysarthria. J Speech Lang Hear Res. 2020 Apr 27;63(4):1106-1114. doi: 10.1044/2020_JSLHR-19-00233. Epub 2020 Apr 17. PMID 32302251